CLINICAL TRIAL: NCT07168837
Title: Letrozole and Cabergoline Versus Letrozole Alone in Ovulation Induction Among PCOS Patients in Assiut Governorate
Brief Title: Letrozole and Cabergoline Versus Letrozole Alone in Ovulation Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Esraa Hamouda Mohammed Ramadan, Resident of Obstetrics & Gynecology, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Letrozole and Cabergoline
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2023-01

CONDITIONS: PCOS (Polycystic Ovary Syndrome)
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Letrozole; Cabergoline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Letrozole with cabergoline) (Active Comparator): About 50 of infertile female with PCOs whom received Letrozole, 5mg daily for 5 days, from day 3 of the cycle up to 7th day for 3 cycles in addition to cabergoline, 0.5 mg weekly for 12 weeks.
  Interventions: Drug: Letrozole tablets
- Group B (Letrozole only) (Active Comparator): About 50 of infertile female with PCOs whom received Letrozole only, 5mg daily for 5 days, from day 3 of the cycle up to 7th day for 3 cycles.
  Interventions: Drug: Letrozole tablets

INTERVENTIONS:
Drug: Letrozole tablets — to compare between Letrozole withncabergoline and letrozole alone in ovulation induction among PCOS female patients.
  Other Names: Cabergoline

SUMMARY:
Polycystic Ovarian Syndrome (PCOS) is the most common endocrine disorders in women of reproductive age. According to the World Health Organization (WHO) estimation revealed over 116 million women (3.4%) are affected by PCOS worldwide.

Owing to the intricacy of this condition, various sets of diagnostic criteria have been initiated for the confirmation of PCOS which are: National Institute of Health, Rotterdam's Criteria, Androgen Excess and PCOS society. The prevalence of PCOS is estimated at about 4 to 21 % when it is diagnosed according to the Rotterdam criteria accounting for 75% of cases with anovulatory infertility.

DETAILED DESCRIPTION:
In women with PCOS, the serum FSH levels are slightly lower during the follicular phase, therefore aromatization of excessive androgens is insufficient, and the follicles will not undergo the final FSH-dependent maturation in a dominant follicle. Furthermore, the serum level of anti-Mullerian hormone (AMH) is elevated. AMH counteracts the FSH-driven aromatase complex activity, so high AMH levels will inhibit granulosa cell conversion of androgens to estrogens and have a detrimental effect on final follicular maturation.

Previous studies showed that 30% of patients with PCOS show a modest rise in prolactin level. Increasing serum prolactin in these patients could be detected in both follicular and luteal phase of the normal and stimulated cycles. Dopamine release from the hypothalamus inhibits prolactin secretion, and it also affects the secretion of gonadotropins. When this inhibitory effect of dopamine is reduced, prolactin secretion will increase in addition to abnormalities in gonadotropins including luteinizing hormones.

Cabergoline which is a dopamine receptor agonist, with higher affinity to dopamine D2 receptors had improved uterine perfusion and achieved a better ovulatory response in PCOS patients, due to its ability to inhibit the vascular endothelial growth factor (VEGF) secretion in luteinized granulosa cells. Other studies concluded that Cabergoline use could normalize androgen level and therefore improve the menstrual irregularity in women with PCOS.

Letrozole is a third-generation aromatase inhibitor. It blocks the conversion of C-19 androgens to C-18 estrogens by competitively inhibiting the enzyme, aromatase (cytochrome P-450), which is an essential step in estrogen biosynthesis in the ovary and other tissues.The subsequent feedback to the hypothalamus containing reduced estrogen levels, triggers a compensatory increase in hypothalamic gonadotropin-releasing hormone (GnRH) secretion, and thus an increased release of pituitary gonadotropins FSH & LH. These gonadotropins subsequently promote growth of the follicles and stimulate ovulation. Letrozole has 99.9% bioavailability after oral administration. It has a single dose terminal half-life of 42 hours.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with PCOS according to Rotterdam criteria (Rotterdam, 2004) as:

  1. Menstrual anomalies like amenorrhea (no cycles in the past 6 months), oligomenorrhoea (cycles lasting longer than 35 days), or long cycles.
  2. Clinical and/or biochemical hyperandrogenism.
  3. Ultrasound (USG) appearance of polycystic ovaries (multiple cysts >12 in number of 2-9 mm size).

     Exclusion Criteria:
* Patient with liver and kidney disease.
* Congenital adrenal hyperplasia.
* Hypothalamic or pituitary cause of amenorrhea.
* Primary hyperprolactinemia.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Identification of Ovulation | One week from drug taking
  Detection of Ovulation among the women whom participated and took the drugs of the study by making Serial ultrasound monitoring started from day 10 of menstrual cycle.

CONTACTS AND LOCATIONS:
Overall Officials: El-Kotb Hasan El-Kotb El-Saeidy, Professor, Study Chair — Obstetrics and Gynecology Department, Faculty of medicine,Al-Azhar University, Assiut.
Locations (1):
- Al-Azhar University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided